CLINICAL TRIAL: NCT05686070
Title: A Multicenter, International, Randomized, Placebo Controlled, Double-blind, Parallel Group and Event Driven Phase 3 Study of the Oral FXIa Inhibitor Asundexian (BAY 2433334) for the Prevention of Ischemic Stroke in Male and Female Participants Aged 18 Years and Older After an Acute Non-cardioembolic Ischemic Stroke or High-risk TIA
Brief Title: A Study to Test Asundexian for Preventing a Stroke Caused by a Clot in Participants After an Acute Ischemic Stroke or After a High-risk Transient Ischemic Attack, a So-called Mini Stroke
Acronym: OCEANIC-STROKE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20604; 2023-503793-20-00 (Other: CTIS (EU)); 2022-001067-27 (EudraCT Number)
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Prevention of Ischemic Stroke; Acute Non-cardioembolic Ischemic Stroke; High-risk Transient Ischemic Attack
MeSH Terms: interventions — asundexian

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Asundexian (Experimental): Participants will receive asundexian.
  Interventions: Drug: Asundexian (BAY2433334)
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asundexian (BAY2433334) — Once daily, oral
  Arms: Asundexian
Drug: Placebo — Placebo to asundexian, once daily, oral
  Arms: Placebo

SUMMARY:
Researchers are looking for a better way to prevent an ischemic stroke which occurs when a blood clot travelled to the brain in people who within the last 72 hours had:

* an acute stroke due to a blood clot that formed outside the heart (acute non-cardioembolic ischemic stroke), or
* TIA/mini-stroke with a high risk of turning into a stroke (high-risk transient ischemic attack), and who are planned to receive standard of care therapy. Acute ischemic strokes or TIA/mini-stroke result from a blocked or reduced blood flow to a part of the brain. They are caused by blood clots that travel to the brain and block the vessels that supply it. If these blood clots form elsewhere than in the heart, the stroke is called non-cardioembolic. People who already had a non-cardioembolic stroke are more likely to have another stroke. This is why they are treated preventively with an antiplatelet therapy, the current standard of care. Antiplatelet medicines prevent platelets, components of blood clotting, from clumping together.

Anticoagulants are another type of medicine that prevents blood clots from forming by interfering with a process known as coagulation (or blood clotting).

The study treatment asundexian is a new type of anticoagulant currently under development to provide further treatment options. Asundexian aims to further improve the standard of care without increasing the risk of bleeding.

The main purpose of this study is to learn whether asundexian works better than placebo at reducing ischemic strokes in participants who recently had a non-cardioembolic ischemic stroke or TIA/mini-stroke when given in addition to standard antiplatelet therapy. A placebo is a treatment that looks like a medicine but does not have any medicine in it.

Another aim is to compare the occurrence of major bleeding events during the study between the asundexian and the placebo group. Major bleedings have a serious or even life-threatening impact on a person's health.

Dependent on the treatment group, the participants will either take asundexian or placebo once a day for at least 3 months up to 31 months.

Approximately every 3 months during the treatment period, either a phone call or a visit to the study site is scheduled on an alternating basis. In addition, one visit before and up to two visits after the treatment period are planned.

During the study, the study team will:

* Check vital signs such as blood pressure and heart rate
* Examine the participants' heart health using an electrocardiogram (ECG)
* Take blood samples
* Ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments. In addition, the participants will be asked to complete a questionnaire on quality of life at certain time points during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years of age
* Acute non-cardioembolic stroke or high-risk TIA
* Systemic or cerebrovascular atherosclerosis or acute non-lacunar infarct

Exclusion Criteria:

* Ischemic stroke ≤ 7 days before the index event
* Index stroke following procedures or strokes due to other rare causes
* History of atrial fibrillation/flutter, left ventricular thrombus, mechanic valve or other cardioembolic source of stroke requiring anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12327 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-10-23 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of ischemic stroke | Up to 31 months
Time to first occurrence of ISTH major bleeding | Up to 31 months
  ISTH=International Society on Thrombosis and Hemostasis

SECONDARY OUTCOMES:
Time to first occurrence of all strokes (ischemic and hemorrhagic) | Up to 31 months
Time to first occurrence of composite of CV death, MI or stroke | Up to 31 months
  CV=Cardiovascular, MI=Myocardial infarction
Time to first occurrence of composite of all-cause mortality, MI or stroke | Up to 31 months
Time to first occurrence of disabling stroke (mRS ≥3 at 90 days) | Up to 31 months
  mRS=Modified Rankin Scale
Time to first occurrence of all-cause mortality | Up to 31 months
Time to first occurrence of transient ischemic attack (TIA) | Up to 31 months
Time to first occurrence of composite of ISTH major or clinically relevant non-major bleeding | Up to 31 months
Time to first occurrence of ISTH clinically relevant non-major bleeding | Up to 31 months
Time to first occurrence of symptomatic intracranial hemorrhage | Up to 31 months
Time to first occurrence of hemorrhagic stroke | Up to 31 months
Time to first occurrence of fatal bleeding | Up to 31 months
Time to first occurrence of minor bleeding | Up to 31 months
Time to first occurrence of composite of ischemic stroke or ISTH major bleeding | Up to 31 months
Time to first occurrence of composite of CV death, all stroke, MI or ISTH major bleeding | Up to 31 months
Time to first occurrence of composite of all-cause mortality, disabling stroke, fatal bleeding, symptomatic intracranial hemorrhage | Up to 31 months
Time to first occurrence of ischemic stroke in the first 90 days | Up to 31 months

CONTACTS AND LOCATIONS:
Locations (741):
- United States (108):
  - Eastern Shore Research Institute, LLC | Fairhope, AL, Fairhope, Alabama
  - Barrow Neurologic Institute - Petznick Stroke Center, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Banner - University Medical Center Tucson - Neurology, Tucson, Arizona
  - University of Arkansas for Medical Sciences - Neurology, Little Rock, Arkansas
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - Long Beach Medical Center - Neurology, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center - Neurology, Los Angeles, California
  - Los Angeles - USC Healthcare Center 2 - Neurology, Los Angeles, California
  - UCLA NeuroTranslational Research Center, Los Angeles, California
  - Hoag Memorial Hospital - Center for Research & Education, Newport Beach, California
  - UCI Medical Center - Neurology, Orange, California
  - San Francisco VA Health Care System, San Francisco, California
  - Cottage Health | Santa Barbara Cottage Hospital - Research Department, Santa Barbara, California
  - The Lundquist Institute - Neurology, Torrance, California
  - St. Vincent's Medical Center - Neurology Clinic, Bridgeport, Connecticut
  - Nuvance Health, Danbury, Connecticut
  - Yale University | School of Medicine - Department of Neurology, New Haven, Connecticut
  - ChristianaCare Health Services | Christiana Hospital - Emergency Medicine Research, Newark, Delaware
  - HCA Florida JFK Hospital - Neurology, Atlantis, Florida
  - Delray Medical Center - Neurology, Boynton Beach, Florida
  - Nova Clinical Research - Blake Medical Center, Bradenton, Florida
  - BayCare Health System | Morton Plant Hospital - Neuroscience Research department, Clearwater, Florida
  - UF Health Neuromedicine Hospital, Gainesville, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - Intercoastal Medical Group | Clinical Research, Sarasota, Florida
  - USF Health South Tampa Center for Advanced Healthcare - Neurology, Tampa, Florida
  - BayCare Health System | Saint Joseph's Hospital - Neurology Department, Tampa, Florida
  - University of Illinois Hospital - Neurology, Chicago, Illinois
  - The University of Chicago Medical Center - Neurology, Chicago, Illinois
  - Loyola University Medical Center - Neurology, Maywood, Illinois
  - Mercyhealth Javon Bea Hospital - Riverside | Neurology Research Department, Rockford, Illinois
  - HSHS St. John's Hospital - Neurology, Springfield, Illinois
  - Baptist Health Lexington, Lexington, Kentucky
  - Ochsner Medical Center - New Orleans - Neurology, New Orleans, Louisiana
  - University of Maryland Medical Center - Neurology Care Center, Baltimore, Maryland
  - Tufts Medical Center - Neurology, Boston, Massachusetts
  - Henry Ford Hospital - Neurology, Detroit, Michigan
  - MSU Health Care Neurology & Ophthalmology, East Lansing, Michigan
  - Trinity Health | Oakland Hospital - Clinical Research Department, Pontiac, Michigan
  - Minneapolis Clinic of Neurology | Golden Valley, MN, Golden Valley, Minnesota
  - Mayo Clinic - Rochester - Neurology, Rochester, Minnesota
  - University Hospital - UMMC - Neurology, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City - Neurology, Kansas City, Missouri
  - Kansas City VA Medical Center - Neurology, Kansas City, Missouri
  - Barnes-Jewish Hospital - Cardiology, St Louis, Missouri
  - Mercy Research - St. Louis, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center - Neurology, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Albany Medical College | Department of Neurology, Albany, New York
  - SUNY Downstate Health Sciences University - Neurology, Brooklyn, New York
  - NYU Langone Hospital Brooklyn - Neurology, Brooklyn, New York
  - Mount Sinai Brooklyn - Neurology, Brooklyn, New York
  - Trinity Medical Western New York | Trinity Vascular & Endovascular Center - Research Department, Buffalo, New York
  - Neuroscience Institute at Great Neck, Great Neck, New York
  - Westchester Medical Center, Hawthorne, New York
  - The Neurological Institute - Columbia University Irving Medical Center, New York, New York
  - Mount Sinai Hospital - Stroke Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Rochester General Hospital, Rochester, New York
  - Mission Hospital | Neurology, Asheville, North Carolina
  - Duke Neurological Disorders Clinic - Clinic 1L, Durham, North Carolina
  - Guilford Neurologic Research Partners, LLC., Greensboro, North Carolina
  - ECU Health Medical Center - Neurology, Greenville, North Carolina
  - North Carolina Heart & Vascular (Capital Heart), Raleigh, North Carolina
  - Novant Health Forsyth Medical Center - Neurology, Winston-Salem, North Carolina
  - Atrium Health Wake Forest Baptist | Medical Center - Neurology Department, Winston-Salem, North Carolina
  - Cleveland Clinic - Neurology, Cleveland, Ohio
  - Ohio State University Wexner Medical Center - Neurology, Columbus, Ohio
  - OhioHealth Neuroscience Center at Riverside, Columbus, Ohio
  - Wright State University | Boonshoft School of Medicine - WSU and Premier Health Clinical Trials Research Alliance, Dayton, Ohio
  - Kettering Health Main Campus - Neurology, Kettering, Ohio
  - Mercy Health - St. Rita's Medical Center - Neurology, Lima, Ohio
  - ProMedica | ProMedica Toledo Hospital - Neuro/Stroke Research Department, Toledo, Ohio
  - Mercy Health St. Vincent Medical Center - Neurology, Toledo, Ohio
  - Mercy Health St. Elizabeth Youngstown Hospital - Neurology, Youngstown, Ohio
  - OU Health University of Oklahoma Med Center - Neurology, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - OHSU Hospital - Neurology, Portland, Oregon
  - LVH Neurology - 1250 Cedar Crest, Allentown, Pennsylvania
  - University of Pittsburgh Medical Center, Hamot | Clinical Trials and Research, Erie, Pennsylvania
  - UPMC Harrisburg - Cardiology, Harrisburg, Pennsylvania
  - Penn State Milton S. Hershey Medical Center - Neurology, Hershey, Pennsylvania
  - Lancaster General Health Neuroscience Institute, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania - Neurology, Philadelphia, Pennsylvania
  - Jefferson Hospital for Neuroscience, Philadelphia, Pennsylvania
  - Lewis Katz School of Medicine at Temple University | Neurology, Philadelphia, Pennsylvania
  - Jefferson Einstein Philadelphia Hospital - Neurology, Philadelphia, Pennsylvania
  - Rhode Island Hospital - Neurology, Providence, Rhode Island
  - MUSC Health Neurology at Rutledge Tower, Charleston, South Carolina
  - Prisma Health Greenville Memorial Hospital - Comprehensive Stroke Center, Greenville, South Carolina
  - Erlanger Neurology, Chattanooga, Tennessee
  - The University of Tennessee Medical Center - Main Campus - Neurology, Knoxville, Tennessee
  - Baptist Memorial Hospital East - Cardiology, Memphis, Tennessee
  - Baylor University Medical Center at Dallas - Neurology, Dallas, Texas
  - James W. Aston Ambulatory Care Center - Neurology, Dallas, Texas
  - Doctors Hospital at Renaissance - Neurology, Edinburg, Texas
  - Texas Health Harris Methodist Hospital - Fort Worth - Neurology, Fort Worth, Texas
  - Houston Methodist Neurological Institute, Houston, Texas
  - UTHealth Houston Neurosciences Neurology - Texas Medical Center, Houston, Texas
  - Neurology Consultants of Dallas - Plano, Plano, Texas
  - UT Health San Antonio - Medical Arts & Research Center - Neurology, San Antonio, Texas
  - Baylor Scott & White Medical Center - Temple - Neurology, Temple, Texas
  - Intermountain Cardiovascular Research Department, Murray, Utah
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah
  - Neurological Associates - Henrico, Henrico, Virginia
  - Marshall University Medical Center - Neurology, Huntington, West Virginia
  - Froedtert Hospital - Neurology, Milwaukee, Wisconsin
- Argentina (15):
  - Clinica IMA, Adrogué, Buenos Aires
  - Hospital General de Agudos JM Ramos Mejia | Neurologia Vascular - Enfermedades Cerebrovasculares, Buenos Aires (Capital Federal), Buenos Aires
  - Hospital General de Agudos Dr. Ignacio Pirovano | Infectology, Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Hospital Italiano de La Plata | Clinical Research Department, La Plata, Buenos Aires
  - Policlinico Lomas | Neurology Department, Lomas de Zamora, Buenos Aires
  - Hospital Privado de Comunidad | Clinical Research Department, Mar del Plata, Buenos Aires
  - Galeno | Sanatorio de la Trinidad Mitre - Neurology Department, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Fleni | Sede Belgrano - Neurology Department, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Complejo Medico Policial Churruca Visca | Neurology department, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Instituto Universitario Hospital Italiano de Buenos Aires | Hospital Italiano de Buenos Aires - Neurology Department, Ciudad Autonoma de Buenos Aire, Ciudad Auton. de Buenos Aires
  - Grupo Gamma | Hospital Privado de Rosario, Neurology Department, Rosario, Santa Fe Province
  - Sanatorio Parque | Departamento de Neurologia, Rosario, Santa Fe Province
  - Centro Estudios Médicos e Invest. Clínicas "Dr. N. Quirno", Buenos Aires
  - Sanatorio Allende | Departamento de Investigación Clínica, Córdoba
  - San Bernardo Hospital | Neurology Department, Salta
- Australia (25):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Blacktown Hospital, Blacktown, New South Wales
  - South Western Sydney Local Health District | Liverpool Hospital - Stroke and Neurovascular Department, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal Prince Alfred Hospital, Newtown, New South Wales
  - Prince of Wales Hospital NSW, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Nepean Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital Australia, Brisbane, Queensland
  - Redcliffe District Hospital, Redcliffe, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Grampians Health Ballarat, Ballarat, Victoria
  - Eastern Health Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Western Health Neuroscience Research Unit, St Albans, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (12):
  - Landesklinikum Moedling | Abteilung für Neurologie, Mödling, Lower Austria
  - Universitätsklinikum St. Pölten, Sankt Pölten, Lower Austria
  - Kardinal Schwarzenberg Klinikum, Schwarzach im Pongau, Salzburg
  - Universitaetsklinikum Graz | Abteilung für Neurologie, Graz, Styria
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Kepler Universitaetsklinikum GmbH- Med Campus III - Klinik fuer Neurologie 2, Linz, Upper Austria
  - Barmherzige Brueder Linz | Neurologie, Linz, Upper Austria
  - LKH Feldkirch / Neurologie, Feldkirch, Vorarlberg
  - Barmherzige Brueder Wien | Abt. fuer Neurologie, Vienna
  - AKH Wien | Univ. Klinik fuer Neurologie, Vienna
  - Klinik Ottakring | Neurologische Abteilung, Vienna
  - Klinik Floridsdorf | Abt. f. Neurologie, Vienna
- Belgium (12):
  - Jessa Hospital | Neurology Department, Hasselt, Limburg
  - Hôpital Erasme/Erasmus Ziekenhuis - Neurology department, Anderlecht
  - AZ Sint-Jan Brugge | Neurology, Bruges
  - UZ Brussel, Brussels
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - UZ Gent, Ghent
  - AZ Groeninge Campus Kennedylaan - Neurology department, Kortrijk
  - UZ Leuven - Neurology department, Leuven
  - CHC MontLégia Neurology Department, Liège
  - Kust, Ommeland en Meetjesland (KOM) Network | AZ Damiaan - Neurology Department, Ostend
  - Vitaz | Sint-Niklaas Hospital - Cardiology Department, Sint-Niklaas
  - Clinique de l'Europe, Uccle
- Brazil (17):
  - Hospital Geral de Fortaleza, Fortaleza, Ceará
  - Hospital Estadual Central Vitoria - Fundação INOVA - ES, Espirito Santo, Espírito Santo
  - Centro de Pesquisas do Hospital Bahia, Salvador, Estado de Bahia
  - Hospital Universitário UFMS, Campo Grande, Mato Grosso do Sul
  - Hospital da Universidade Federal de Minas Gerais, Belo Horizonte, Minas Gerais
  - Hospital Madre Tereza, Belo Horizonte, Minas Gerais
  - Hospital das Clinicas da Universidade Federal do Paraná, Curitiba, Paraná
  - Hospital Moinhos de Vento-Centro Clínico, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre | Clinical Research Center - Surgery Research Center, Porto Alegre, Rio Grande do Sul
  - Clinica Neurologica e Neurocirurgica de Joinville Ltda, Joinville, Santa Catarina
  - Hospital das Clínicas de Botucatu - UNESP Botucatu, Botucatu, São Paulo
  - Sociedade Matonense de Benemerência, Matão, São Paulo
  - Fundação Facu. Reg de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Nove de Julho, São Paulo, São Paulo
  - L'Dor - Instituto de Ensino e Pesquisa, Rio de Janeiro
  - Science Valley Research Institute, São Paulo
  - Unifesp/Epm, São Paulo
- Bulgaria (18):
  - Multispecialty Hospital for Active Treatment St. Ivan Rilski - 2003 | Neurological Department, Dupnitsa
  - Multiprofile Hospital for Active Treatment Haskovo AD | Department of Nervous Diseases, Haskovo
  - Multiprofile Hospital for Active Treatment Pazardzhik, Pazardzhik
  - Military Medical Academy | Multiprofile Hospital for Active Treatment Pleven - Neurology Department, Pleven
  - University Multiprofile Hospital for Active Treatment Dr Georgi Stranski Pleven | Department of Neurology, Pleven
  - Multiprofile Hospital for Active Treatment Saint Panteleimon Hospital | Neurology Department, Plovdiv
  - University Multiprofile Hospital for Active Treatment Pulmed | Neurology Department, Plovdiv
  - University Multispecialty Hospital for Active Treatment 'Kanev' JSC | Department of General and Vascular Neurology, Rousse
  - Military Medical Academy | Multiprofile Hospital for Active Treatment Sofia - Clinic of Neurological Diseases, Sofia
  - Second Multi-profile Hospital for Active Treatment - Sofia | Clinic of Neurology, Sofia
  - Multiprofile Hospital for Active Treatment National Cardiology Hospital | Clinic for Neurological Diseases, Sofia
  - Acibadem City Clinic University Multiprofile Hospital For Active Treatment Tokuda - Department of Neurology and Sleep Medicine, Sofia
  - University Hospital for Active Treatment Tsaritsa Joanna - ISUL | Neurology Department, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N. I. Pirogov EAD - Department of Nervous Diseases, Sofia
  - Multiprofile Hospital for Active Treatment Neurology and Psychiatry St. Naum | Intensive Treatment of Nervous System Disorders, Sofia
  - University Multiprofile Hospital for Active Treatment Sofiamed | Neurology Department, Sofia
  - University Hospital for Active Treatment St. Anna | Neurology Department, Sofia
  - MHAT Sveta Marina EAD, Varna
- Canada (22):
  - University of Calgary | Foothills Medical Centre - Department of Clinical Neurosciences - Stroke Clinical Trials Group, Calgary, Alberta
  - University of Alberta Hospital - Canada, Edmonton, Alberta
  - Center For Neurologic Research, Lethbridge, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Vancouver General Hospital / Vancouver Stroke Program, Vancouver, British Columbia
  - Winnepeg Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Complex, Halifax, Nova Scotia
  - Health Sciences North Research Institute | Sudbury, Canada, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston Health Sciences Centre (KGH Site), Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital | The Ottawa Hospital Research Institute - Neurology - Ottawa Stroke Program, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Unity Health Toronto | St. Michael's Hospital - Stroke Research, Toronto, Ontario
  - CIUSSS Saguenay Lac-St-Jean, Chicoutimi, Quebec
  - CHUM - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Center - Neurology Department, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Québec-Hôpital de l'Enfant-Jésus, Québec, Quebec
  - CIUSSS de l'Estrie-CHUS, Hopital Fleurimont, Sherbrooke, Quebec
  - University of Saskatchewan, Royal University Hospital, Saskatoon, Saskatchewan
- China (59):
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Foshan First People's Hospital, Foshan, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou Overseas Chinese Hospital, Guangzhou, Guangdong
  - People's Hospital of Liuzhou City, Liuchow, Guangxi
  - Hainan General Hospital, Haikou, Hainan
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hengshui Harrison International Peace Hospital, Hengshui, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Tangshan people's Hospital, Tangshan, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - Daqing People's Hospital, Daqing, Heilongjiang
  - 1st Affiliated Hospital of Henan Science and Technology Univ, Luoyang, Henan
  - Luoyang Third People's Hospital, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - The Third Affiliated Hospital of Xinxiang Medical university, Xinxiang, Henan
  - The Central Hospital of Wuhan, Tongji Medl Collg Huazhong..., Wuhan, Hubei
  - Puai Hospital,Tongji Medical College, Huazhong Univ Sci&Tech, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - 1st Affiliated Hospital of Nanhua University, Hengyang, Hunan
  - Baogang hospital, Baotou, Inner Mongolia
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - The Affiliated Huaian No.1 People's Hospi of NJ Medical Unv., Huai'an, Jiangsu
  - Affiliated Hospital of Jiangsu University, JiangSu, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical university, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Wuxi No.2 People's Hospital, Wuxi, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Baoji Central Hospital, Baoji, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Yan'an University Xianyang Hospital, Xianyang, Shaanxi
  - Qilu Hosp., Shandong Univ., Jinan, Shandong
  - Jining No.1 people's Hospital, Jining, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - People's Hospital of Deyang City, Deyang, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang Univ. School of Medicine, Hangzhou, Zhejiang
  - Hwa Mei Hospital, University of Chinese Academy Sciences, Ningbo, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Xuanwu Hospital Capital Medical University, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Huashan Hospital, Fudan University, Shanghai
  - Yangpu Hospital, Tongji University, Shanghai
  - Tianjin People's Hospital, Tianjin
  - Tianjin Huanhu Hospital, Tianjin
- Colombia (16):
  - Hospital Alma Mater de Antioquia, Medellín, Antioquia
  - Hospital General de Medellin, Medellín, Antioquia
  - Promotora Médica Las Américas S.A.- Clinica Las Americas, Medellín, Antioquia
  - Sociedad Médica Rionegro SOMER S.A., Rionegro, Antioquia
  - Clínica de la Costa SAS, Baranquilla, Atlántico
  - Fundación Hospital Universidad del Norte, Soledad, Atlántico
  - Hospital Universitario Mayor-MÉDERI, Bogotá, Bogota D.C.
  - Clínica Universidad de la sabana, Chía, Cundinamarca
  - Cardiomet Cequin Sas, Armenia, Quindío Department
  - Clínica Imbanaco S.A.S, Cali, Valle del Cauca Department
  - Fundación Valle de Lili, Cali
  - Fundación Oftalmológica de Santander Carlos Ardila Lule, Florida Blanca
  - Fundación Cardiovascular de Colombia, Floridablabca
  - Hospital San Vicente Fundación, Medellín
  - Clínica Medellín, Medellín
  - Clinica Cardio VID, Medellín
- Czechia (15):
  - Fakultni nemocnice u sv. Anny - I.neurologicka klinika, Brno
  - Nemocnice Chomutov, o.z., Chomutov
  - Nemocnice Ceske Budejovice, a.s. - Department of neurology, České Budějovice
  - Karvinska hornicka nemocnice a.s. - Neurologicke oddeleni, Fryštát
  - Nemocnice Jihlava - Neurologicke oddeleni, Jihlava
  - Krajska nemocnice Liberec - neurologicke oddeleni, Liberec
  - Fakultni nemocnice Ostrava - Neurologicka klinika, Ostrava - Poruba
  - Nemocnice AGEL Ostrava-Vítkovice a. s. - Neurologické oddelení, Ostrava - Vitkovice
  - Nemocnice Pardubickeho Kraje, as - Neurologická klinika, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady - Neurologicka klinika, Prague
  - Fakultni Thomayerova Nemocnice - neurology department, Prague
  - Ustredni vojenska nemocnice Praha, Prague
  - Nemocnice na Homolce - Neurology Department, Praha 5-Motol
  - Krajská Zdravotní, Masarykova nemocnice Ústí nad Labem - Neurologické oddelení, Ústí nad Labem
  - Krajská nemocnice T. Bati - Neurologické oddelení, Zlín
- Denmark (8):
  - Aalborg Universitetshospital - Neurologisk afdeling, Aalborg
  - Aarhus Universitetshospital, Neurologisk Afdeling, Aarhus N
  - Rigshospitalet Glostrup - Hjerne og Nervesygdomme, Glostrup Municipality
  - Herlev Hospital - Hjerne og Nervesygdomme, Herlev
  - Regionshospitalet Gødstrup - Neurologi, Herning
  - Lillebælt Sygehus Kolding - Hjerne og Nervesygdomme, Kolding
  - Bispebjerg Hospital - Neurologisk afdeling, København NV
  - Odense Universitetshospital - Neurologisk afdeling, Odense C
- Finland (5):
  - HUS, Meilahden sairaala, Helsinki
  - Pohjois-Karjalan sairaanhoitopiiri, Joensuu
  - Kuopion yliopistollinen sairaala, Kuopio
  - Tampere University Hospital, Tampereen yliopistollinen sairaala (TAYS), Tampere
  - Turun yliopistollinen keskussairaala, Turku
- France (29):
  - HCL - Hopital Louis Pradel - Service de Neurologie, Bron, Auvergne-Rhône-Alpes
  - AP-HM - Hopital de la Timone - Service de Neurologie, Marseille, Bouches-du-Rhône
  - CHU Strasbourg - Hopital Hautepierre - Service Neurologie, Strasbourg, Grand Est
  - CHRU Besancon - Hopital Jean Minjoz - Service neurologie, Besançon
  - Hopital Pellegrin _ Soins Intensifs Unite Neurovasculaire, Bordeaux
  - Centre Hospitalier Boulogne sur Mer - Neurologie, Boulogne-sur-Mer
  - CHU de Brest - Hopital La Cavale Blanche, Brest
  - CH Sud Francilien, Neurologie, Corbeil-Essonnes
  - CHU Dijon - Hopital Francois Mitterand - Service neurologie generale vasculaire et degenerative, Dijon
  - Hopital Raymond-Poincare _ Service de Neurologie, Garches
  - Assistance Publique Hopitaux de Paris (AP-HP) - Hopital Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier - Le Mans _ Service de Neurologie, Le Mans
  - Hopital Salengro _ Service de Neurologie et Pathologie Neurovasculaire, Lille
  - GHICL - Hopital Saint-Philibert, Lomme
  - CHRU Nancy - Hopital central - Service de neurologie, Nancy
  - CHU de Nice - Hopital Pasteur - Unite Neuro Vasculaire, Nice
  - Hopital Caremeau _ Service de Neurologie, Nîmes
  - Hopital de la Pitie-Salpetriere _ Service des Urgences Cerebro-Vasculaires, Paris
  - Centre hospitalier Sainte Anne, Paris
  - APHP Hopital Bichat Claude Bernard - Service de Neurologie, Paris
  - APHP - Hopital Fondation Adolphe De Rothschild - Service de Neurologie, Paris
  - AP-HP - Hopital Lariboisiere, Paris
  - CHU de Reims - Hopital de la Maison Blanche - Service de Neurologie, Reims
  - CHU Rennes - Hopital Pontchaillou - Service de neurologie, Rennes
  - CHU de Nantes - Hopital Laennec - Unite neurovasculaire, Saint-Herblain
  - Hopital Foch - Service de Neurologie, Suresnes
  - Hopital instruction des Armees Sainte Anne, Toulon
  - CHU Toulouse - Hopital Pierre Paul Riquet PURPAN, Toulouse
  - CHRU de Tours - Hôpital Bretonneau - Service de neurologie, Tours
- Germany (28):
  - Universitätsklinikum Freiburg / Neurologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Heidelberg / Neurologie, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Ulm/Neurologische Klinik, Ulm, Baden-Wurttemberg
  - Rhön-Klinikum Campus Bad Neustadt/Neurologie, Bad Neustadt an der Saale, Bavaria
  - Universitätsklinikum Erlangen/Neurologie, Erlangen, Bavaria
  - Universitätsklinikum Frankfurt / Neurologie, Frankfurt am Main, Hesse
  - Universität Gießen-Marburg, Standort Gießen/Neurologie, Giessen, Hesse
  - Universitätsmedizin Göttingen/ Neurologie, Göttingen, Lower Saxony
  - Medizinische Hochschule Hannover/Neurologie, Hanover, Lower Saxony
  - Universitätsmedizin Greifswald/Neurologie, Greifswald, Mecklenburg-Vorpommern
  - UniKlinikum Aachen/Neurologie, Aachen, North Rhine-Westphalia
  - Uniklinik Bonn / Neurologie, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf / Neurologie, Düsseldorf, North Rhine-Westphalia
  - Marien Hospital Düsseldorf / Neurologie, Düsseldorf, North Rhine-Westphalia
  - Alfried Krupp Krankenhaus Rüttenscheid /Neurologie, Essen, North Rhine-Westphalia
  - GFO KlinikTroisdorf/Neurologie, Troisdorf, North Rhine-Westphalia
  - Johannes Gutenberg-Universität Mainz - Neurologie, Mainz, Rhineland-Palatinate
  - Städtisches Klinikum Dresden / Neurologie, Dresden, Saxony
  - Universitätsklinikum Dresden/Neurologie, Dresden, Saxony
  - Universitätsklinik Leipzig /Neurologie, Leipzig, Saxony
  - Universitätsklinikum Halle (Saale)/Neurologie, Halle, Saxony-Anhalt
  - Klinikum Altenburger Land / Studienzentrum Neurologie, Altenburg, Thuringia
  - SRH Wald-Klinikum Gera gGmbH, Bad Langensalza, Thuringia
  - Uniklinik Jena/ Neurologie, Jena, Thuringia
  - Vivantes Klinikum Neukölln / Neurologie mit Stroke Unit, Berlin
  - Asklepios Klinik Wandsbek/Neurologie, Hamburg
  - Asklepios Klinik Barmbek/ Neurologie, Hamburg
  - Asklepios Klinik Altona Hamburg / Neurologie, Hamburg
- Greece (17):
  - University General Hospital Of Alexandroupoli- Department of Neurology, Alexandroupoli
  - General Hospital Of Athens Korgialenio Benakio H.R.C.- Department of Neurology, Ampelokipoi Athens
  - Evaggelismos Hospital-Department of Neurology, Athens
  - Naval Hospital of Athens-Department of Neurology, Athens
  - 401 General Military Hospital Of Athens- Department of Neurology, Athens
  - General Hospital Of Athens G Gennimatas- Department of Neurology, Athens
  - Eginitio Hospital-1st Department of Neurology, Athens
  - University General Hospital Attikon-2nd Department of Neurology, Athens
  - General Hospital Of Thessaloniki Papageorgiou-3rd Department of Internal Medicine, Efkarpia
  - University General Hospital of Heraklion - Department of Neurology, Heraklion
  - University General Hospital Of Ioannina-Department of Neurology, Ioannina
  - University General Hospital of Larissa-Department of Neurology, Larissa
  - General University Hospital Of Patras-Department of Neurology, Pátrai
  - Metropolitan Hospital- Stroke Unit, Piraeus
  - University General Hospital Of Thessaloniki Ahepa-2nd Department of Neurology, Thessaloniki
  - University General Hospital Of Thessaloniki Ahepa-1st Department of Neurology, Thessaloniki
  - Geniko Nosokomeio Thessalonikis George Papanikolaou-3rd Department of Neurology, Thessaloniki
- Hungary (16):
  - Bajai Szent Rokus Korhaz, Baja
  - Semmelweis Egyetem, Altalanos Orvostudomanyi Kar, Neurologiai Klinika, Budapest
  - Budapesti Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Eszak-Pesti Centrumkorhaz-Honvedkorhaz, Budapest
  - Semmelweis Egyetem Idegsebeszeti es Neurointervencios Klinika, Budapest
  - Budapesti Jahn Ferenc Del-pesti Korhaz es Rendelointezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont Neurologiai Klinika, Debrecen
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz, Győr
  - Kistarcsai Flor Ferenc Korhaz, Kistarcsa
  - Szent Damján Görögkatolikus Kórház - Neurologiai es Stroke Osztaly, Kisvárda
  - Nagykanizsai Kanizsai Dorottya Korhaz, Nagykanizsa
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Soproni Erzsebet Oktato Korhaz es Rehabilitacios Intezet, Sopron
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Orvostudomanyi Kar Szent-Gyorgyi Albert Klinikai Kozpont Neurologiai Klinika, Szeged
  - Zala Varmegyei Szent Rafael Korhaz, Zalaegerszeg
- India (12):
  - Lalitha Super Specialities Hospital, Guntur, Andhra Pradesh
  - Government General Hospital, Guntur, Guntur, Andhra Pradesh
  - Zydus Hospital, Ahmedabad, Gujarat
  - Aster MIMS Hospital, Kozhikode, Kozhikode, Kerala
  - Sree Chitra Tirunal Institute for Medical Sciences and Technology, Thiruvananthapuram, Kerala
  - Yashoda Hospital, Hyderabad, Telangana
  - K.G. Hospital, Coimbatore
  - Artemis Hospitals, Gūrgaon
  - Shree Krishna Hospital, Karamsad
  - All India Institute of Medical Sciences (AIIMS) - New Delhi, New Delhi
  - Government Medical College - Thiruvanathapuram, Thiruvananthapuram
  - Christian Medical College & Hospital (CMCH) - Vellore, Vellore
- Israel (15):
  - Assuta Ashdod Public Hospital (R.A), Ashdod
  - Barzilai Medical Center | Neurology Department, Ashkelon
  - Clalit Health | Soroka Medical Center - Internal Medicine Department, Beersheba
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Corporation, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Edith Wolfson Medical Center | Internal Medicine Department, Holon
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center | Beilinson Hospital - Internal Medicine C Department, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Health Corporation of the Ziv Medical Center (R.A.), Safed
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin
- Italy (22):
  - Azienda Sanitaria Locale Avezzano Sulmona L'Aquila - Ospedale SS. Filippo e Nicola - Neurologia, Avezzano, Abruzzo
  - Azienda Ospedaliero Universitaria Delle Marche - Clinica Neurologica, Torrette, Ancona
  - ASL Della Provincia Di Lecce_Ospedale Vito Fazzi - Neurologia, Lecce, Apulia
  - Azienda Ospedaliera Di Rilievo Nazionale Antonio Cardarelli - Neurologia, Napoli, Campania
  - A.O.U San Giovanni Di Dio E Ruggi d'Aragona - Neurologia e Stroke Unit, Salerno, Campania
  - Azienda Unita Sanitaria Locale Di Bologna_ Ospedale Maggiore Pizzardi - Neurologia, Bologna, Emilia-Romagna
  - AUSL della Romagna_Ospedale Bufalini - Neurologia, Cesena, Emilia-Romagna
  - Azienda Ospedaliero Universitaria Parma - SC Percorso Stroke Care, Parma, Emilia-Romagna
  - ASU Friuli Centrale_Ospedale "Santa Maria della Misericordia" - Neuroscienze, Udine, Friuli Venezia Giulia
  - Azienda Ospedaliera Policlinico Universitario Tor Vergata - UOSD Stroke Unit, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Neurologia, Rome, Lazio
  - Azienda Sociosanitaria Ligure 2_Ospedale Santa Corona - Neurologia Ponente, Pietra Ligure, Liguria
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII - Neurologia, Bergamo, Lombardy
  - Ospedale San Raffaele s.r.l. - Neurologia, Milan, Lombardy
  - Azienda Ospedaliera Universitaria Gaetano Martino Messina - Stroke Unit, Messina, Sicily
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello - Neurologia e Stroke Unit, Palermo, Sicily
  - Careggi University Hospital - Stroke Unit, Florence, Tuscany
  - Azienda Ospedaliera Universitaria Senese - Stroke unit, Siena, Tuscany
  - A.O. di Perugia_Hospital Santa Maria della Misericordia - S.S. Stroke Unit, Perugia, Umbria
  - IRCCS Ospedale Sacro Cuore Don Calabria - Neurologia, Negrar, Veneto
  - Azienda Ospedaliera Universitaria Integrata Verona_Borgo Trento - Neurologia A, Verona, Veneto
  - Azienda Sanitaria Locale Citta Di Torino - Ospedale San Giovanni Bosco - Neurologia 2, Torino
- Japan (66):
  - Nagoya Ekisaikai Hospital, Nagoya, Aichi-ken
  - Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Tosei General Hospital, Seto, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - National Hospital Organization Toyohashi Medical Center, Toyohashi, Aichi-ken
  - Kimitsu Chuo Hospital, Kisarazu, Chiba
  - Toho University Sakura Medical Center, Sakura, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Steel Memorial Yawata Hospital, Kitakyushu, Fukuoka
  - Southern Tohoku Medical Clinic, Kōriyama, Fukushima
  - Japanese Red Cross Takayama Hospital, Takayama, Gifu
  - Maebashi Red Cross Hospital, Maebashi, Gunma
  - Mazda Motor Corporation Mazda Hospital, Aki-gun, Hiroshima
  - Hiroshima General Hospital, Hatsukaichi, Hiroshima
  - Higashihiroshima Medical Center, Higashihiroshima, Hiroshima
  - Japanese Red Cross Asahikawa Hospital, Asahikawa, Hokkaido
  - Hakodate Shintoshi Hospital, Hakodate, Hokkaido
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Ohnishi Neurological Center, Akashi, Hyōgo
  - Hyogo Prefectural HarimaHimeji General Medical Center, Himeji, Hyōgo
  - Eishokai Yoshida Hospital, Kobe, Hyōgo
  - JA Toride Medical Center, Toride, Ibaraki
  - Tsuchiura Kyodo General Hospital, Tsuchiura, Ibaraki
  - Japan Organization of Occupational Health and Safety Kagawa Rosai Hospital, Marugame, Kagawa-ken
  - Takamatsu Red Cross Hospital, Takamatsu, Kagawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Nippon Medical School Musashikosugi Hospital, Kawasaki-shi, Kanagawa
  - Seisho Hospital, Odawara, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital, Yokohama, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - Uji-Tokushukai Medical Center, Uji, Kyoto
  - Kohnan Hospital, Sendai, Miyagi
  - Japan Culture and Welfare Federation of Agricultural Cooperatives | Hokushin General Hospital, Nakano, Nagano
  - Japanese Red Cross Society Suwa Hospital, Suwa, Nagano
  - National Hospital Organization Beppu Medical Center, Beppu, Oita Prefecture
  - Japanese Red Cross Okayama Hospital, Okayama, Okayama-ken
  - Nozaki Tokushukai Hospital, Daitō, Osaka
  - Kotobuki Social Medical Corporation Tominaga Hospital, Osaka, Osaka
  - Osaka Saiseikai Senri Hospital, Suita, Osaka
  - National Hospital Organization Ureshino Medical Center, Ureshino, Saga-ken
  - Hamamatsu Rosai Hospital, Hamamatsu, Shizuoka
  - National Hospital Organization Tokyo Medical Center, Meguro-ku, Tokyo
  - Mishuku Hospital, Meguro-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Sumida-ku, Tokyo
  - National Hospital Organization Disaster Medical Center, Tachikawa, Tokyo
  - Minamiwakayama Medical Center, Tanabe, Wakayama
  - JCHO Shimonoseki Medical Center, Shimonoseki, Yamaguchi
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Saiseikai Fukuoka General Hospital, Fukuoka
  - Social Medical Corporation the Chiyukai foundation Fukuoka Wajiro Hospital, Fukuoka
  - Fukuoka Neurosurgical Hospital, Fukuoka
  - Kyushu Central Hospital, Fukuoka
  - Hiroshima City North Medical Center Asa Citizens Hospital, Hiroshima
  - Japanese Red Cross Kochi Hospital, Kochi
  - Kumamoto City Hospital, Kumamoto
  - Koseikai Takeda Hospital, Kyoto
  - Ijinkai Takeda General Hospital, Kyoto
  - Nagano Municipal Hospital, Nagano
  - CMIC HealthCare Institute Co. Ltd. | Local IAA OCGMC - Okayama City Civic Hospital - Clinical Trial Centre, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Shizuoka City Shizuoka Hospital, Shizuoka
  - Shizuoka City Shimizu Hospital, Shizuoka
  - Wakayama Medical University Hospital, Wakayama
- Kazakhstan (3):
  - Multiprofile regional hospital, Aktobe
  - City Clinical Hospital No7 - Stroke Unit, Almaty
  - Multidisciplinary City Hospital No1 - Stroke Unit, Astana
- Latvia (5):
  - Daugavpils Regional Hospital, Daugavpils
  - Jekabpils Regional Hospital, Jēkabpils
  - Rezekne Hospital, Rēzekne
  - P. Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital "Gailezers", Riga
- Lithuania (5):
  - Alytus County S. Kudirka Hospital, Alytus
  - Hospital of LT University of Health Sciences Kaunas Clinics, Kaunas
  - Siauliai Republican hospital, Šiauliai
  - Republican Vilnius University Hospital, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Malaysia (9):
  - Hospital Raja Perempuan Zainab II, Kelantan
  - Hospital Universiti Sains Malaysia, Kelantan
  - Queen Elizabeth Hospital Malaysia, Kota Kinabalu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Sultan Abdul Aziz Shah, Kuala Selangor
  - Hospital Seberang Jaya, Pulau Pinang
  - Sarawak General Hospital, Sarawak
  - Hospital Sultanah Nur Zahirah Medical Department, Terengganu
- Netherlands (11):
  - Catharina Hospital | Neurology Outpatient Clinic, Eindhoven, North Brabant
  - Jeroen Bosch Ziekenhuis | Department of Neurology, 's-Hertogenbosch
  - OLVG | Location West - Neurology Department, Amsterdam
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Zuyderland Medical Centre | Sittard-Geleen - Neurology Department, Heerlen
  - St. Antonius Hospital | Nieuwegein - Neurology Department - Stroke Unit, Nieuwegein
  - Maasstad Ziekenhuis | Neurology Department, Rotterdam
  - HagaZiekenhuis | Department of Neurology, The Hague
  - University Medical Center (UMC) Utrecht | Neurology and Neurosurgery Department, Utrecht
  - Isala Zwolle | Neurology Department, Zwolle
- Norway (6):
  - Ålesund sykehus Nevrologisk poliklinikk, Ålesund
  - Haukeland Universitetssykehus Nevrologisk Avdeling, Bergen
  - Östfold Hospital Trust Fredrikstad, Grålum
  - Akershus Universitetssykehus - Nevrologisk Avdeling, Lørenskog
  - Molde sykehus Nevrologisk avdeling, Molde
  - OUS Ullevål Neurology Department, Oslo
- Poland (13):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Uniwersytecki Nr 2 im. J. Bizela, Bydgoszcz
  - Copernicus PL, M.Kopernik Hospital, Gdansk
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni im. sw. Jana Pawla II, Grodzisk Mazowiecki
  - Górnoslaskie Centrum Medyczne im. prof. Leszka Gieca Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Szpital Specjalistyczny im. Rydygiera, Krakow
  - Samodzielny Publiczny Szpital Kliniczny nr 4, Lublin
  - Wojewodzki Szpital Specjalistyczny im. sw. Jadwigi w Opolu, Opole
  - SP Szpital Kliniczny nr 1 PUM im. Prof. T. Sokolowskiego, Szczecin
  - Szpital Wolski im. dr Anny Gostynskiej SPZOZ, Warsaw
  - Instytut Psychiatrii i Neurologii w Warszawie, Warsaw
  - Wojskowy Instytut Medyczny Panstwowy Instytut Badawczy, Warsaw
- Portugal (12):
  - Hospital Professor Doutor Fernando Fonseca | Neurology Department, Amadora, Lisbon District
  - Hospital Pedro Hispano | Clinical Research Center, Matosinhos Municipality, Porto District
  - Unidade Local de Saude Almada-Seixal | Hospital Garcia de Orta - Research Department, Almada, Setúbal District
  - Centro Hospitalar e Universitario de Coimbra | Hospitais da Universidade de Coimbra - Neurology Department, Coimbra
  - Centro Hospitalar Universitario do Algarve | Faro - Ensino, Inovacao e Investigacao - Centro de Investigacao e Documentacao, Faro
  - Centro Hospitalar de Leiria | Santo Andre Hospital - Research Center, Leiria
  - Unidade Local De Saúde De Lisboa Ocidental E.P.E., Lisbon
  - Luz Saude | Hospital da Luz Lisboa - Centro de Investigacao Clinica, Lisbon
  - CHULN - Hospital Santa Maria, Lisbon
  - BlueClinical | Centro Hospitalar Baixo Vouga - Unidade Aveiro - Gabinete de Ensaios Clinicos, Lisbon
  - Centro Hospitalar Universitario do Porto | Servico de Investigacao Clinica, Porto
  - Centro Hospitalar Universitario de Sao Joao | Polo Porto - Centro de Investigacao e Ensaios Clinicos, Porto
- Slovakia (16):
  - Univerzitna nemocnica Bratislava, Nemocnica Stare Mesto, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica ak. L.Derera, Bratislava
  - Dolnooravska nemocnica s poliklinikou L. Nadasi Jegeho, Dolný Kubín
  - Nemocnica AGEL Komarno s.r.o., Komárno
  - Vseobecna nemocnica s poliklinikou Levoca, a.s., Levoča
  - Liptovska nemocnica s poliklinikou MUDr. Ivana Stodolu, Liptovský Mikuláš
  - Univerzitna nemocnica Martin, Martin
  - Fakultna nemocnica Nitra, Nitra
  - Fakultna nemocnica s poliklinikou J.A. Reimana, Prešov
  - Penta Hospitals | Rimavska Sobota Hospital - Neurology Department, Rimavská Sobota
  - Fakultna nemocnica AGEL Skalica, a.s., Skalica
  - Nemocnica s poliklinikou Spisska Nova Ves a.s., Spišská Nová Ves
  - Fakultna nemocnica Trnava, Trnava
  - ProCare Svet Zdravia | Vranov nad Toplou Hospital - Neurology Department, Vranou Nad Toplou
  - Nemocnica AGEL Ziar nad Hronom a Banska Stiavnica s.r.o., Žiar nad Hronom
- South Korea (21):
  - Kyungpook National University Hospital, Daegu, Daegu Gwang''yeogsi
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggido
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Severance Hospital, Yonsei University Health System-Neurology instead of Cardiology, Seoul, Seoul Teugbyeolsi
  - University of Ulsan College of Medicine - Asan Medical Center (AMC) - Cardiology Department, Seoul, Seoul Teugbyeolsi
  - Kyung Hee University Medical Center, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Eulji University Hospital, Daejeon
  - Chonnam National University Hospital, Dong-gu, Gwangju
  - Inha University Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - SoonChunHyang University Seoul Hospital, Seoul
  - Samsung Medical Center-Neurology instead of Cardiology, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
- Spain (25):
  - University Hospital of A Coruna | Neurology Department - Stroke, No-Cardioembolic-Tia, A Coruña, A Coruña
  - Hospital Clinico Universitario de Santiago de Compostela | Neurology Department - Stroke, No-Cardioembolic-Tia, Santiago de Compostela, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Rey Juan Carlos - Neurologia, Móstoles, Madrid
  - Hospital Alvaro Cunqueiro | Neurology Department - Stroke, No-Cardioembolic-Tia, Babio - Beade, Pontevedra
  - IIS Biobizkaia Health Research Institute | Hospital de Cruces - Neurology Department - Stroke, No-Cardioembolic-Tia, Barakaldo, Vizcaya
  - Hospital General Universitario De Albacete - Neurologia, Albacete
  - Hospital de la Santa Creu i Sant Pau | Neurology Department - Stroke, No-Cardioembolic-Tia, Barcelona
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Universitari De Girona Doctor Josep Trueta - Neurologia, Girona
  - Hospital Universitario De Leon - Neurologia, León
  - Hospital Universitari Arnau De Vilanova De La Gerencia Territorial De Lleida - Neurologia, Lleida
  - COMPLEJO HOSPITALARIO RUBER JUAN BRAVO - Neurología, Madrid
  - Hospital Universitario de La Princesa | Neurology Department, Madrid
  - H Gregorio Marañon|Neurology|STROKE|NO-CARDIOEMBOLIC-TIA, Madrid
  - Hospital Universitario Ramon Y Cajal - Neurologia, Madrid
  - Hospital Universitario 12 de Octubre | Neurology Department - Stroke, No-Cardioembolic-Tia, Madrid
  - Hospital Universitario La Paz | Neurology Department - Stroke, No-Cardioembolic-Tia, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca | Neurology Department - Stroke, Murcia
  - Hospital Universitario Virgen De La Macarena - Neurologia, Seville
  - Hospital Universitario Virgen Del Rocio S.L. - Neurologia, Seville
  - Hospital Universitari Joan XXIII De Tarragona - Neurologia, Tarragona
  - Hospital Clinico Universitario de Valencia | Neurology Department, Valencia
  - Hospital Universitario Y Politecnico La Fe - Neurologia, Valencia
  - Hospital Clinico Universitario De Valladolid - Neurologia, Valladolid
- Sweden (8):
  - Danderyds sjukhus, Danderyd
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skånes Universitetssjukhus, Lund
  - Östersunds Sjukhus, Östersund
  - Södersjukhuset AB, Stockholm
  - Karolinska University Hospital, Huddinge Neuroradiology, Stockholm
  - Karolinska University Hospital, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Switzerland (9):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Hôpital Cantonal Universitaire de Genève, Geneva, Canton of Geneva
  - Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Ospedale regionale di Lugano, Lugano, Canton Ticino
  - Inselspital Universitätsspital Bern, Bern
  - Hospital Cantonal Fribourg, Villars-sur-Glâne
  - NeuroZentrum Hirslanden, Zurich
- Taiwan (24):
  - China Medical University Hospital Hsin-Chu Branch, Zhubei, Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - Far Eastern Memorial Hospital Neurology, New Taipei City, Taipei
  - En Chu Kong Hospital, New Taipei City, Taipei
  - Fu Jen Catholic University Hospital, New Taipei City, Taipei
  - MacKay Memorial Hospital Tamsui Branch, New Taipei City, Taipei
  - Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital, Hsin-Chu Branch, Hsinchu
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Chang Gung Memorial Hospital Keelung, Keelung
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi-Mei Medical Center, Liouyine, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- Turkey (Türkiye) (21):
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Health Ministry Of Türkiye Republic Ankara Bilkent City Hospital, Ankara
  - Akdeniz Universitesi Tip Fakultesi Hastanesi, Antalya
  - Firat Universitesi Tip Fakultesi, Elâzığ
  - Eskisehir Osmangazi Universitesi Tip Fakultesi, Eskişehir
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Bakirkoy Prof Dr Mazhar Osman Ruh Sagligi ve Sinir Hast. EAH, Istanbul
  - Istanbul Sultan 2. Abdulhamid Han Egitim ve Arastirma Has., Istanbul
  - Kartal Dr Lutfi Kirdar Sehir Hastanesi, Istanbul
  - Marmara Uni. Tip Fak. Pendik EAH Noroloji, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Saglik Bilimleri Universitesi Izmir Tepecik EAH, Izmir
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Selcuk University Faculty of Medicine, Konya
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi Hastanesi, Konya
  - Samsun Egitim Arastirma Hastanesi, Samsun
  - Ondokuz Mayis Uni Tip Fakultesi, Samsun
  - Cumhuriyet Universitesi Tip Fakultesi, Sivas
- United Kingdom (16):
  - Southampton General Hospital, Southampton, Hampshire
  - East Kent Hospitals University NHS Foundation Trust | Kent and Canterbury Hospital - Stroke Unit, Canterbury, Kent
  - St George's University Hospitals NHS Foundation Trust | St George's Hospital | Neurology Department, Kogarah, London
  - Northern Care Alliance NHS Foundation Trust | Salford Royal Hospital - Clinical Research Facility, Salford, Manchester
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust | Royal Victoria Infirmary - Acute Stroke Unit, Newcastle upon Tyne, Tyne and Wear
  - South Tyneside and Sunderland NHS Foundation Trust | Sunderland Royal Hospital - Acute Stroke Unit, Sunderland, Tyne and Wear
  - Leeds Teaching Hospitals NHS Trust | Leeds General Infirmary - Cardiology, Leeds, West Yorkshire
  - University Hospitals of Derby and Burton NHS Foundation Trust | Royal Derby Hospital - Cardiology, Derby
  - Edinburgh Royal Infirmary, Edinburgh
  - Royal Devon University Healthcare NHS Foundation Trust | Royal Devon and Exeter Hospital - Stroke Unit, Exeter
  - NHS Greater Glasgow and Clyde | Glasgow Royal Infirmary |Glasgow Research Facility - Cardiology, Glasgow
  - Liverpool University Hospitals NHS Foundation Trust | Aintree University Hospital - Stroke Unit, Liverpool
  - King's College Hospital NHS Foundation Trust | King's College Hospital - Academic Neuroscience Centre, London
  - Charing Cross Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Sharma M, Dong Q, Hirano T, Kasner SE, Saver J, Masjuan J, Demchuk AM, Cordonnier C, Bereczki D, Tsivgoulis G, Veltkamp R, Staikov I, Bae HJ, Campbell BCV, Zini A, Lee IH, Ameriso S, Kovar M, Mikulik R, Lemmens R, Ferro JM, Robinson T, Christensen H, Ozturk S, Leker RR, Turcani P, Slowik A, Amaya P, Hoo FK, De Marchis GM, Knoflach M, Sylaja PN, Putaala J, Coutinho JM, Worp HBV, Miglane E, Matijosaitis V, Lindgren AG, Silva GS, Sandset EC, Turuspekova ST, Joundi RA, Schulze K, Shestakovska O, Gilbride J, Bangdiwala SI, Xu L, Muehlhofer E, Colorado P, Mundl H, Keller L, Shoamanesh A. Rationale, design and baseline characteristics of participants in the OCEANIC-STROKE trial of FXIa inhibition for secondary stroke prevention. Eur Stroke J. 2026 Jan 1;11(1):aakaf017. doi: 10.1093/esj/aakaf017. PMID 41614533
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/20604